CLINICAL TRIAL: NCT05274750
Title: A Randomised, Double-blind, Parallel Group Phase III Study to Assess the Efficacy and Safety of 100 mg SC Depemokimab in Patients With Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) - ANCHOR-1 (depemokimAb iN CHrOnic Rhinosinusitis)
Brief Title: Efficacy and Safety of Depemokimab (GSK3511294) in Participants With Chronic Rhinosinusitis With Nasal Polyps
Acronym: ANCHOR-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 217095; 2021-005037-16 (EudraCT Number)
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Nasal Polyps
Keywords: Depemokimab; GSK3511294; Chronic rhinosinusitis; Verbal response scale; Asthma Control Questionnaire; Lund Mackay computed tomography; Nasal polyps score; Nasal endoscopy
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Intervention Model Description: Participants will receive either depemokimab (GSK3511294) or placebo during the study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This will be a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Depemokimab (Experimental): Participants received a 100 milligram (mg) dose of depemokimab SC injection once every 26 weeks (week 0 and week 26) over a treatment period of 52 weeks. Participants were to be maintained on their existing baseline maintenance for Chronic Rhinosinusitis with Nasal Polyps (CRSwNP) standard of care (SOC) treatment throughout the study.
  Interventions: Biological: Depemokimab (GSK3511294)
- Placebo (Placebo Comparator): Participants received placebo SC injection once every 26 weeks (week 0 and week 26) over a treatment period of 52 weeks. Participants were to be maintained on their existing baseline maintenance for CRSwNP SOC treatment throughout the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Depemokimab (GSK3511294) — Depemokimab (GSK3511294) was administered using a pre- filled syringe.
  Arms: Depemokimab
Drug: Placebo — Placebo was administered as normal saline using a pre-filled syringe.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of depemokimab (GSK3511294) in participants with Chronic rhinosinusitis with nasal polyps (CRSwNP).

ELIGIBILITY:
Inclusion criteria:

* Participants with 18 years of age and older inclusive, at the time of signing the informed consent.
* Endoscopic bilateral NP score of at least 5 out of a maximum score of 8 (with a minimum score of 2 in each nasal cavity) assessed by the investigator.
* Participants who have had at least one of the following at Visit 1: Previous nasal surgery for the removal of NP; have used at least three consecutive days of systemic corticosteroids in the previous 2 years for the treatment of NP; medically unsuitable or intolerant to systemic corticosteroid.
* Participants (except for those in Japan) must be on daily treatment with intranasal corticosteroids (INCS) (including intranasal liquid steroid wash/douching) for at least the 8 weeks immediately prior to screening.
* Participants presenting with severe NP symptoms defined as symptoms of nasal congestion/blockade/obstruction with moderate or severe severity and loss of smell or rhinorrhea (runny nose) based on clinical assessment by the investigator.
* Presence of symptoms of chronic rhinosinusitis as described by at least 2 different symptoms for at least 12 weeks prior to Visit 1, one of which should be either nasal blockage/obstruction/congestion or nasal discharge (anterior/posterior nasal drip), plus facial pain/pressure and/or reduction or loss of smell.
* Male or eligible female participants.

Exclusion criteria:

Exclusion criteria:

* As a result of medical interview, physical examination, or screening investigation the physician responsible considers the participant unfit for the study.
* Cystic fibrosis.
* Antrochoanal polyps.
* Nasal cavity tumor (malignant or benign).
* Fungal rhinosinusitis.
* Severe nasal septal deviation occluding one nostril preventing full assessment of nasal polyps in both nostrils
* Participants who had a sino-nasal or sinus surgery changing the lateral wall structure of the nose making impossible the evaluation of nasal polyp score.
* Acute sinusitis or upper respiratory tract infection (URTI) at screening or in 2 weeks prior to screening.
* Ongoing rhinitis medicamentosa (rebound or chemical induced rhinitis).
* Participants who have had an asthma exacerbation requiring admission to hospital within 4 weeks of screening.
* Participants who have undergone any intranasal and/or sinus surgery (for example [e.g.], polypectomy, balloon dilatation or nasal stent insertion) within 6 months prior to Visit 1; nasal biopsy prior to Visit 1 for diagnostic purposes only is excepted.
* Participants where NP surgery is contraindicated in the opinion of the Investigator.
* Participants with other conditions that could lead to elevated eosinophils such as hyper-eosinophilic syndromes including (but not limited to) Eosinophilic granulomatosis with polyangiitis (EGPA) (formerly known as Churg-Strauss Syndrome) or Eosinophilic Esophagitis.
* Participants with a known, pre-existing parasitic infestation within 6 months prior to Visit 1.
* A known immunodeficiency (e.g. human immunodeficiency virus [HIV]), other than that explained by the use of corticosteroids (CSs) taken as therapy for asthma.
* A current malignancy or previous history of cancer in remission for less than 12 months prior to screening.
* Liver Disease: Alanine aminotransferase (ALT) >2 times Upper limit of normal (ULN); Total bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin less than [<]35 percent [%]); Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice.
* Participants who have known, pre-existing, clinically significant cardiac, endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, hematological or any other system abnormalities that are uncontrolled with standard treatment.
* Participants with current diagnosis of vasculitis. Participants with high clinical suspicion of vasculitis at screening will be evaluated and current vasculitis must be excluded prior to enrollment.
* Hypersensitivity: Participants with allergy/intolerance to the excipients of depemokimab (GSK3511294) in a monoclonal antibody, or biologic.
* Participants that, according to the investigator's medical judgment, are likely to have active Coronavirus Disease-2019 (COVID-19) infection must be excluded. Participants with known COVID-19 positive contacts within the past 14 days must be excluded for at least 14 days following the exposure during which the participant should remain symptom-free. Reported smell/ taste complications from COVID-19 must be used as exclusion.
* Participants that have been exposed to ionizing radiation in excess of 10 millisievert (mSv) above background over the previous 3-year period as a result of occupational exposure or previous participation in research studies.
* Previously participated in any study with mepolizumab, reslizumab, or benralizumab and received study intervention (including placebo) within 12 months prior to Visit 1.
* Women who are pregnant or lactating or are planning on becoming pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (90):
- United States (25):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Buena Park, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Temecula, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Richmond, Virginia
- Argentina (7):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Florida
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, Mar del Plata
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Rosario
- GSK Investigational Site, Ghent, Belgium
- Canada (5):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- China (10):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Dongguan
  - GSK Investigational Site, Jingzhou
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Qingdao
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Taiyuan
  - GSK Investigational Site, Wenzhou
  - GSK Investigational Site, Wuhan
  - GSK Investigational Site, Yantai
- France (11):
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, La Roche-sur-Yon
  - GSK Investigational Site, La Rochelle
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Pontoise
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Valenciennes
- Germany (8):
  - GSK Investigational Site, Bonn
  - GSK Investigational Site, Dortmund
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Düsseldorf
  - GSK Investigational Site, Marburg
  - GSK Investigational Site, München
  - GSK Investigational Site, Münster
  - GSK Investigational Site, Wiesbaden
- Japan (11):
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Leiden
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Jerez de la Frontera
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Zaragoza
- United Kingdom (3):
  - GSK Investigational Site, Great Yarmouth
  - GSK Investigational Site, Stevenage
  - GSK Investigational Site, Wigan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

REFERENCES:
- [Background] Gevaert P, Cornet M, Mullol J, De Corso E, Keles Turel N, Desrosiers M, et al. . ANCHOR-1/-2 primary data including pooled analysis ms. Lancet. PMID: 40037388 DOI: 10.1016/S0140-6736(25)00197-7
- [Derived] Jackson DJ, Bourdin A, Blackorby A, Leslie A, Vichiendilokkul A, Howarth P, Karkoszka N, Fujieda S, Cornet M. Safety and Tolerability of Twice-Yearly Depemokimab in Patients with Asthma and Chronic Rhinosinusitis with Nasal Polyps: Pooled Results from SWIFT-1/-2 and ANCHOR-1/-2. Adv Ther. 2025 Dec 29. doi: 10.1007/s12325-025-03457-4. Online ahead of print. PMID 41461999
- [Derived] Gevaert P, Desrosiers M, Cornet M, Mullol J, De Corso E, Keles Turel N, Maspero J, Fujieda S, Zhang L, Sousa AR, Woods SJ, Davis AM, Schalkwijk S, Edwards D, Ranganathan P, Follows R, Marshall C, Han JK; ANCHOR-1 and ANCHOR-2 trial investigators. Efficacy and safety of twice per year depemokimab in chronic rhinosinusitis with nasal polyps (ANCHOR-1 and ANCHOR-2): phase 3, randomised, double-blind, parallel trials. Lancet. 2025 Mar 15;405(10482):911-926. doi: 10.1016/S0140-6736(25)00197-7. Epub 2025 Mar 1. PMID 40037388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 276 participants were randomized to the study. Of which 271 participants were included in the Full analysis set (FAS) population. The FAS included all randomized participants who received at least 1 dose of study intervention excluding 4 participants from 1 site with Good clinical practice (GCP)/data integrity issues. One participant was randomized in error and did not receive any study drug.
Pre-assignment Details: A total of 276 participants were enrolled in the study.
Period: Overall Study
Arm/Group | Depemokimab | Placebo
Started | 143 | 133
Full Analysis Population | 143 | 128
Completed | 128 | 115
Not Completed | 15 | 18
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 10 | 9
Not completed — GCP Violation | 0 | 4
Not completed — Randomized, not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) population included all randomized participants who received at least one dose of study intervention excluding participants from 1 site with GCP violation. Participants were analyzed according to the intervention they were allocated at randomization.
Groups:
- Depemokimab: Participants received a 100 mg dose of depemokimab SC injection once every 26 weeks (week 0 and week 26) over a treatment period of 52 weeks. Participants were to be maintained on their existing baseline maintenance for CRSwNP SOC treatment throughout the study.
- Total: Total of all reporting groups
Arm/Group | Depemokimab | Placebo | Total
Number analyzed (Participants) | 143 | 128 | 271
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 54.1 (13.37) | 52.9 (13.49) | 53.5 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 38 | 83
  Male | 98 | 90 | 188
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 37 | 30 | 67
  BLACK OR AFRICAN AMERICAN | 4 | 2 | 6
  WHITE | 97 | 88 | 185
  UNKNOWN | 1 | 4 | 5
  MISSING | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Endoscopic Nasal Polyps (NP) Score at Week 52 (Centrally Read)
Description: Total endoscopic nasal polyps (NP) score evaluated the size and extent of nasal polyps via endoscopy. The assessments were performed by central video image recordings of nasal endoscopy. The right and left nostrils were scored from 0 to 4 (0 = No polyps; 1 = Small polyps in the middle meatus not reaching below the inferior border of the middle concha; 2 = Polyps reaching below the lower border of the middle turbinate; 3 = Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle concha; and 4 = Large polyps causing complete obstruction of the inferior meatus). The scores were graded based on NP size, recorded as sum of the right and left nostril scores and ranges from 0 (no polyps) to 8 (large polyps), calculated by summing the scores [0 to 4] in each nostril; with higher scores indicating worse status. Baseline was defined as Day 1 value. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and at Week 52
Population: The FAS included all randomized participants who received at least one dose of study intervention excluding participants from 1 site with GCP violation. The overall number of participants analyzed represents only those participants available at the specified time points and evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Depemokimab | Placebo
Number analyzed (Participants) | 139 | 127
Scores on a Scale | -0.6 (0.14) | 0.2 (0.15)
Statistical Analysis 1: Comparison: Depemokimab vs Placebo; To assess the efficacy of depemokimab 100mg SC + SoC compared to placebo + SoC at Week 52 in participants with a diagnosis of CRSwNP; Test type: Other — Analysis performed using a repeated measures model with covariates of treatment group, baseline score, log(e) baseline blood eosinophil count, region, previous surgery for nasal polyps, visit, visit by baseline, and visit by treatment group; p < 0.001, Mixed Models Analysis; Difference in Least Square Means = -0.7, 95% CI 2-sided [-1.1 to -0.3]

2. Primary Outcome: Change From Baseline in Mean Nasal Obstruction Score Using Verbal Response Scale From Week 49 Through to Week 52
Description: This endpoint evaluated the change from baseline in the mean nasal obstruction score using a Verbal Response Scale (VRS) from Week 49 through to Week 52. Participants used a VRS to rate nasal obstruction severity, with scores averaged over the specified period to assess treatment impact on nasal obstruction symptoms. Participants were asked to indicate the severity of nasal obstruction at their worst over the last 24 hours using a 4-point VRS, with options of no symptoms, mild symptoms, moderate symptoms, and severe symptoms. This was scored on a scale ranging from 0 (no symptoms) to 3 (severe symptoms), with higher scores indicating worse status. The average of daily scores in 4-weekly intervals were calculated and data are presented for Weeks 49-52. Baseline was defined as the average score from 28 days of electronic diary (eDiary) data collected prior to Day 1. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and from Week 49 to Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Depemokimab | Placebo
Number analyzed (Participants) | 142 | 128
Scores on a Scale | -0.76 (0.079) | -0.53 (0.083)
Statistical Analysis 1: Comparison: Depemokimab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.047, Mixed Models Analysis; Difference in Least Square Means = -0.23, 95% CI 2-sided [-0.46 to 0.00]

3. Secondary Outcome: Change From Baseline in Mean Symptom Score for Rhinorrhea (Runny Nose) Using Verbal Response Scale From Week 49 Through to Week 52
Description: Participants were asked to indicate the severity of rhinorrhea (runny nose) at their worst over the last 24 hours using a 4-point VRS, with options of no symptoms, mild symptoms, moderate symptoms, and severe symptoms. This was scored on a scale ranging from 0 (no symptoms) to 3 (severe symptoms). Higher scores indicate the worse status. The average of daily scores in 4-weekly intervals were calculated and data are presented for Weeks 49-52. Baseline was defined as the average score from 28 days of eDiary data collected prior to Day 1. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and from Week 49 to Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Depemokimab | Placebo
Number analyzed (Participants) | 142 | 128
Scores on a Scale | -0.71 (0.084) | -0.49 (0.087)
Statistical Analysis 1: Comparison: Depemokimab vs Placebo; To assess the efficacy of depemokimab 100mg SC + SoC compared to placebo + SoC at Week 49 to Week 52 in participants with a diagnosis of CRSwNP; Test type: Other — Analysis performed using a repeated measures model with covariates of treatment group, baseline score, log(e) baseline blood eosinophil count, region, previous surgery for nasal polyps, visit, visit by baseline, and visit by treatment group. If the hierarchy is broken, subsequent endpoints will be evaluated for nominal significance in a descriptive manner, using a 5 percent (%) reference level; p = 0.074, Mixed Models Analysis; Difference in Least Square Means = -0.22, 95% CI 2-sided [-0.46 to 0.02]

4. Secondary Outcome: Change From Baseline in Mean Symptom Score for Loss of Smell Using Verbal Response Scale From Week 49 Through to Week 52
Description: Participants were asked to indicate the severity of loss of smell at their worst over the last 24 hours using a 4-point VRS, with options of no symptoms, mild symptoms, moderate symptoms, and severe symptoms. This was scored on a scale ranging from 0 (no symptoms) to 3 (severe symptoms). Higher score indicates worse status. The average of daily scores in 4-weekly intervals were calculated and data are presented for Weeks 49-52. Baseline was defined as the average score from 28 days of eDiary data collected prior to Day 1. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and from Week 49 to Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Depemokimab | Placebo
Number analyzed (Participants) | 142 | 128
Scores on a Scale | -0.48 (0.069) | -0.29 (0.072)
Statistical Analysis 1: Comparison: Depemokimab vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other — Analysis performed using a repeated measures model with covariates of treatment group, baseline score, log(e) baseline blood eosinophil count, region, previous surgery for nasal polyps, visit, visit by baseline, and visit by treatment group. If the hierarchy is broken, subsequent endpoints will be evaluated for nominal significance in a descriptive manner, using a 5% reference level; p = 0.055, Mixed Models Analysis; Difference in Least Square Means = -0.19, 95% CI 2-sided [-0.39 to 0.00]

5. Secondary Outcome: Change From Baseline in Lund Mackay Computerized Tomography (CT) Score at Week 52
Description: The LMK CT scoring system is based on CT imaging of the sinuses with points given for degree of opacification: 0 =normal, 1 = partial opacification, 2 = total opacification. These points were applied to the maxillary, anterior ethmoid, posterior ethmoid, sphenoid, frontal sinus on each side (right and left). The osteomeatal complex (OC) is graded as 0 = not occluded, or 2 = occluded. The range for the total LMK CT score is therefore 0 (normal) to 24 (total opacification) when summed across both sides with higher scores indicating more severe disease. Baseline was defined as Day 1 value. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Depemokimab | Placebo
Number analyzed (Participants) | 127 | 119
Scores on a Scale | -2.8 (0.45) | -0.8 (0.46)
Statistical Analysis 1: Comparison: Depemokimab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Analysis performed using an analysis of covariance model (ANCOVA) with covariates of treatment group, baseline score, log(e) baseline blood eosinophil count, region and previous surgery for nasal polyps. If the hierarchy is broken, subsequent endpoints will be evaluated for nominal significance in a descriptive manner, using a 5% reference level; p = 0.002, ANCOVA; Difference in Least Square Means = -2.0, 95% CI 2-sided [-3.3 to -0.8]

6. Secondary Outcome: Change From Baseline in Sino-nasal Outcome Test (SNOT)-22 Total Score at Week 52
Description: Sino-nasal outcome test-22 is a 22-item measure of disease specific health related quality of life (HRQoL). Participants were asked to rate the severity of their condition on each of the 22 items over the previous 2 weeks using a 6-point rating scale of 0-5 including: 0 = Not present/no problem; 1 = Very mild problem; 2 = Mild or slight problem; 3 = Moderate problem; 4 = Severe problem; 5 = Problem as "bad as it can be". The scores for each question were summed up to derive the total score range for the SNOT-22 was from 0 (high quality of life) to 110 (worst quality of life), where higher scores indicate worse quality of life. Baseline was defined as Day 1 value. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and at Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Depemokimab | Placebo
Number analyzed (Participants) | 139 | 125
Scores on a Scale | -13.3 (2.96) | -6.5 (3.08)
Statistical Analysis 1: Comparison: Depemokimab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.113, Mixed Models Analysis; Difference in Least Square Means = -6.8, 95% CI 2-sided [-15.2 to 1.6]

7. Secondary Outcome: Change From Baseline in Mean Nasal Obstruction Score (Verbal Response Scale) From Week 21 Through to Week 24
Description: Participants were asked to indicate the severity of nasal obstruction at its worst over the previous 24 hours using a 4-point VRS. The response options were no symptoms, mild symptoms, moderate symptoms, and severe symptoms, scored on a scale ranging from 0 (no symptoms) to 3 (severe symptoms). Higher scores indicate more severe status. The average of daily scores in 4-weekly intervals were calculated and data are presented for Weeks 21-24. Baseline was defined as the average score from 28 days of eDiary data collected prior to Day 1. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and from Week 21 to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Depemokimab | Placebo
Number analyzed (Participants) | 142 | 128
Scores on a Scale | -0.74 (0.071) | -0.57 (0.074)
Statistical Analysis 1: Comparison: Depemokimab vs Placebo; To assess the efficacy of depemokimab 100mg SC + SoC compared to placebo + SoC at Week 21 to Week 24 in participants with a diagnosis of CRSwNP; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.094, Mixed Models Analysis; Difference in Least Square Means = -0.17, 95% CI 2-sided [-0.37 to 0.03]

8. Secondary Outcome: Change From Baseline in Total Endoscopic Nasal Polyps Score at Week 26
Description: as for outcome 1
Time Frame: Baseline (Day 1) and at Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Depemokimab | Placebo
Number analyzed (Participants) | 139 | 127
Scores on a Scale | -0.6 (0.13) | 0.1 (0.13)
Statistical Analysis 1: Comparison: Depemokimab vs Placebo; To assess the efficacy of depemokimab 100mg SC + SoC compared to placebo + SoC at Week 26 in participants with a diagnosis of CRSwNP; Test type: Other — [test comment as in outcome 4, analysis 1]; p < 0.001, Mixed Models Analysis; Difference in Least Square Means = -0.8, 95% CI 2-sided [-1.1 to -0.4]

9. Secondary Outcome: Percentage of Participants Requiring First Nasal Surgery (Actual or Entry on Waiting List) or Disease-Modulating Medication for Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) Up to Week 52
Description: Nasal polyp surgery is defined as any procedure involving instruments resulting in incision and removal of tissue from the nasal cavity (for example polypectomy). Time to first nasal polyp surgery (actual or entry on waiting list) or disease-modulating medication for CRSwNP up to Week 52 was assessed in a pre-specified pooled analysis across replicate studies 217095 (NCT05274750) and 218079 (NCT05281523). The percentage of participants with nasal surgery or disease-modulating medication for CRSwNP and corresponding 95% CI have been presented, calculated using the Kaplan-Meier method.
Time Frame: Up to Week 52
Population: For pooled studies of 217095 (NCT05274750) and 218079 (NCT05281523), the analysis was performed on the FAS population. The FAS included all randomized participants who received at least 1 dose of study treatment excluding participants from 1 site for 217095 and 2 sites for 218079 respectively with GCP violation. Participants were analyzed according to the treatment they were allocated at randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pooled Depemokimab: This reporting arm contains the pooled population of treated participants from the clinical trial groups "Depemokimab" study intervention from protocol 217095 and protocol 218079. Participants received a 100 mg dose of depemokimab SC injection once every 26 weeks (week 0 and week 26). Participants were to be maintained on their existing baseline maintenance CRSwNP SOC treatment throughout the study.
- Pooled Placebo: This reporting arm contains the pooled population of participants from the clinical trial groups "Placebo" study intervention from protocol 217095 and protocol 218079. Participants received a Placebo SC injection once every 26 weeks (week 0 and week 26). Participants were to be maintained on their existing baseline maintenance CRSwNP SOC treatment throughout the study.
Arm/Group | Pooled Depemokimab | Pooled Placebo
Number analyzed (Participants) | 272 | 256
Percentage of participants | 15.0 [11.3 to 19.9] | 21.9 [17.2 to 27.7]
Statistical Analysis 1: Comparison: Pooled Depemokimab vs Pooled Placebo; To assess the efficacy of depemokimab 100mg SC + SoC compared to placebo + SoC at Week 52 in participants with a diagnosis of CRSwNP (pooled analysis); Test type: Other — Cox Proportional Hazards Model with covariates of treatment, baseline total endoscopic nasal polyps score, baseline nasal obstruction score (VRS), log(e) baseline blood eosinophil count, region, study and previous surgery for nasal polyps. The covariate for study is removed for the individual-study analyses. If the hierarchy is broken, subsequent endpoints will be evaluated for nominal significance in a descriptive manner, using a 5% reference level; p = 0.128, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.735, 95% CI 2-sided [0.495 to 1.092]

10. Secondary Outcome: Percentage of Participants Requiring First Nasal Surgery (Actual) or Disease-Modulating Medication for CRSwNP up to Week 52
Description: Nasal polyp surgery is defined as any procedure involving instruments resulting in incision and removal of tissue from the nasal cavity (for example polypectomy).Time to first nasal polyp surgery (actual) or disease-modulating medication for CRSwNP up to week 52 was assessed in a pre-specified pooled analysis across replicate studies 217095 (NCT05274750) and 218079 (NCT05281523). The percentage of participants with nasal surgery or disease-modulating medication for CRSwNP and corresponding 95% CI have been presented, calculated using the Kaplan-Meier method.
Time Frame: Up to Week 52
Population: For pooled studies of 217095 (NCT05274750) and 218079 (NCT05281523), the analysis was performed on the FAS population. The FAS included all randomized participants who took at least 1 dose of study treatment excluding participants from 1 site for 217095 and 2 sites for 218079 respectively with GCP violation. Participants were analyzed according to the treatment they were allocated at randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pooled Depemokimab | Pooled Placebo
Number analyzed (Participants) | 272 | 256
Percentage of participants | 12.2 [8.8 to 16.8] | 16.7 [12.6 to 22.0]
Statistical Analysis 1: Comparison: Pooled Depemokimab vs Pooled Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.146, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.713, 95% CI 2-sided [0.453 to 1.124]

11. Secondary Outcome: Percentage of Participants Requiring at Least One Course of Systemic Corticosteroids or Disease-Modulating Medication for CRSwNP or Nasal Surgery (Actual) During the Week 52 Treatment Period
Description: The percentage of participants requiring at least 1 course of systemic corticosteroids (CS) or disease-modulating medication for CRSwNP or nasal surgery (actual) during the Week 52 treatment period was assessed in a pre-specified pooled analysis across replicate studies 217095 (NCT05274750) and 218079 (NCT05281523). Percentage of participants with nasal surgery or course of systemic CS for CRSwNP have been presented.
Time Frame: Up to Week 52
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Pooled Depemokimab | Pooled Placebo
Number analyzed (Participants) | 272 | 256
Percentage of participants | 26 | 36
Statistical Analysis 1: Comparison: Pooled Depemokimab vs Pooled Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Other — Logistic regression with covariates of treatment, number of courses of systemic CS in 12 months prior to screening for NP (0, 1, >1), log(e) baseline blood eosinophil count, baseline total endoscopic NP score, baseline nasal obstruction score (VRS), region, study and previous surgery for NPs. The study covariate is removed for individual study analyses. If the hierarchy is broken, subsequent endpoints will be evaluated for nominal significance in a descriptive manner, using a 5% reference level; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.40 to 0.86]

12. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-5) Score at Week 52
Description: The ACQ-5 is a five-item questionnaire designed to be self-completed by the participants to assess the most common asthma symptoms. The 5 questions enquired to recall how their asthma had been during the previous week and to respond about the frequency and/or severity of symptoms (nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheezing). The overall ACQ-5 response option is the mean score of all 5 questions representing 0 with no impairment/limitation and 6 as total impairment/ limitation. Higher scores indicated more limitations and lower scores with better asthma control. Impact on asthma control in the subgroup of participants with an ACQ-5 score greater than 0.75 (indicating partially or not well-controlled) at baseline was assessed in a pre-specified pooled analysis across replicate studies 217095 (NCT05274750) and 218079 (NCT05281523). Baseline was defined as Day 1 value. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and at Week 52
Population: For pooled studies of 217095 (NCT05274750) and 218079 (NCT05281523), the analysis was performed on the FAS population. The FAS included all randomized participants who took at least 1 dose of study drug excluding participants from 1 site for 217095 and 2 sites for 218079 respectively with GCP violation. Participants were analyzed according to the treatment they were allocated at randomization. The overall number of participants analyzed signifies participants evaluable for specified time points.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Pooled Depemokimab | Pooled Placebo
Number analyzed (Participants) | 104 | 102
Scores on a Scale | -0.75 (0.182) | 0.00 (0.182)
Statistical Analysis 1: Comparison: Pooled Depemokimab vs Pooled Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Other — The pooled statistical analyses will be performed using a Mixed Models Repeated Measures (MMRM) model with covariates of treatment group, baseline score, log(e) baseline blood eosinophil count, region, previous surgery for nasal polyps, study, visit and interaction terms for visit by baseline score and visit by treatment group. If the hierarchy is broken, subsequent endpoints will be evaluated for nominal significance in a descriptive manner, using a 5% reference level; p = 0.004, Mixed Models Analysis; Hazard Ratio (HR) = -0.75, 95% CI 2-sided [-1.26 to -0.25]

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious adverse events (Non-SAEs) were collected from the start of the study intervention (Day 1) till follow up week 56.
Description: All-cause mortality, SAEs and Non-SAEs were reported for the Safety Population which included all randomized participants who received at least 1 dose of study treatment excluding participants from 1 site with GCP violation. AEs were reported treatment-wise.
Arm/Group | Depemokimab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/128
Serious Adverse Events (participants affected / at risk) | 5/143 | 6/128
Other Adverse Events (participants affected / at risk) | 71/143 | 72/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Depemokimab (N=143) | Placebo (N=128)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Depemokimab (N=143) | Placebo (N=128)
Toothache (Gastrointestinal disorders) | 4 (4) | 4 (4)
Acute sinusitis (Infections and infestations) | 7 (9) | 4 (4)
Bronchitis (Infections and infestations) | 6 (6) | 4 (4)
COVID-19 (Infections and infestations) | 12 (12) | 9 (9)
Gastroenteritis (Infections and infestations) | 2 (2) | 4 (5)
Influenza (Infections and infestations) | 3 (4) | 10 (13)
Nasopharyngitis (Infections and infestations) | 21 (28) | 23 (26)
Sinusitis (Infections and infestations) | 5 (7) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 14 (18) | 14 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 6 (6) | 8 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data do not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT05274750/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT05274750/SAP_001.pdf